CLINICAL TRIAL: NCT06761703
Title: Community Outreach Support and Engagement Using Online Strategies - Decentralized Insights Into Therapy Adoption and Value
Brief Title: A Study to Determine the Feasibility of Online Recruitment of People Using an Anti-Obesity Medication for Weight Loss
Acronym: COSMOS-DIGITAL
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20240163
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Adults Using Anti-Obesity Medications: Adults using the anti-obesity medications, semaglutide and tirzepatide, indicated for weight loss to examine the willingness of patients to engage in a digital study, provide consent, and complete various study-related tasks.
  Interventions: Device: TAP® Micro Select Device (Touch Activated Phlebotomy)

INTERVENTIONS:
Device: TAP® Micro Select Device (Touch Activated Phlebotomy) — The TAP Micro Select device will be used in an investigational capacity by participants for self-collection of whole capillary blood.

SUMMARY:
This observational study is designed to determine the feasibility of recruitment from a digital research community of people using an anti-obesity medication for weight loss to understand willingness to consent to survey research and at home self-blood testing. This study will engage an active community of people using anti-obesity medications, semaglutide and tirzepatide, indicated for weight loss to examine the willingness of participants to engage in a digital study, provide consent, and complete various study-related tasks, including a self-collected capillary blood sample for assay testing and health related surveys.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 80 years of age.
* Living in the United States.
* Consented from the Inspire online platform patient community for COSMOS-DIGITAL.
* Self-Reported current use of, and intention to continue for at least 30 days, one of the following medications for the indications of weight management/obesity:
* Semaglutide (wegovy)
* Tirzepatide (zepbound)

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or participation in a current clinical trial.
* Self-reported sensitivity/allergy to any of the components of the self-draw collection device including stainless steel or elements commonly found in stainless steel.
* Self-reported fear of blood.
* Self-reported circulatory conditions causing difficulty in drawing capillary blood.
* Known history of bleeding diathesis or any coagulation disorder.
* History of skin disorders, abnormal skin integrity or atypical skin health within the areas to be tested in the upper arm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults using the anti-obesity medications, semaglutide and tirzepatide, indicated for weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Self-blood Draw Received by Central Laboratory | 30 days

SECONDARY OUTCOMES:
Percentage of Consented Participants with Complete Self-reported Survey for Medical History | Day 1
Percentage of Consented Participants with Complete Self-reported Survey for Nausea and Nausea Management | Day 1 and Day 30
Percentage of Consented Participants with Complete Self-reported Survey for Patient Reported Outcomes in Obesity | Day 1 and Day 30
Percentage of Consented Participants with Complete Self-reported Survey for Partners in Health (PiH) Questionnaire | Day 1 and Day 30
Percentage of Consented Participants with Complete Self-reported Survey for the Daily Diary | 30 days
  The daily diary will record answers about nausea symptoms.
Percentage of Consented Participants with Complete Self-reported Survey for the Satisfaction Survey | Day 30
  Participants will be asked about their satisfaction with using the device for the self-blood draw.
Percentage of Participants with Sufficient Volume of Blood Collected for Sampling | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- YourBio Health/CRT, Medford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com